CLINICAL TRIAL: NCT03884075
Title: Non-Alcoholic Fatty Liver Disease, the Hepatic Response to Oral Glucose, and the Effect of Semaglutide (NAFLD HEROES)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 190072; 19-DK-0072
Record Dates: First submitted 2019-03-20; First posted 2019-03-21 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09-30

CONDITIONS: Non-Alcoholic Steatohepatitis; Non-Alcoholic Fatty Liver Disease
Keywords: Non-Alcoholic Steatohepatitis (NASH); Steatosis; Caloric Load
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — semaglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: Steatosis (Experimental): Participants with steatosis on baseline biopsy
  Interventions: Drug: Semaglutide
- Arm B: NASH (Experimental): Participants with NASH on baseline biopsy
  Interventions: Drug: Semaglutide
- Arm C: Healthy (No Intervention): Healthy Volunteers

INTERVENTIONS:
Drug: Semaglutide — Semaglutide injection once weekly
  Arms: Arm A: Steatosis; Arm B: NASH

SUMMARY:
Background:

In non-alcoholic fatty liver disease (NAFLD), fat accumulates in the liver and can cause damage. Researchers want to learn what causes the damage NAFLD, and to see if a medication can help.

Objective:

To find out how the liver in people with NAFLD responds to feeding, and how this relates to their response to the drug semaglutide.

Eligibility:

People with NAFLD and healthy volunteers ages 18 and older

Design:

Participants will be screened with:

Medical history

Physical exam

Blood tests

Imaging: A machine will take pictures of the participant s body.

Within 2-8 weeks of enrollment, participants will stay in the clinic for several days. This includes:

Blood, urine, heart, and imaging tests

For NAFLD participants only: A needle-like device will remove a small biopsy of the liver and fatty tissue.

Participants will be alone in a special room for 5 hours. They will breathe through a tube under the nostrils. They will have blood drawn several times.

The baseline visit concludes participation for healthy volunteers but NAFLD participants will contine.

About 6 weeks after discharge, participants will stay in the clinic again and repeat the tests. They will get their first semaglutide dose by injection.

Participants will have visits weeks 1, 2, 4, 8, 12, 16, 20, and 24 of treatment. Visits include blood tests.

Participants will inject semaglutide once a week at home.

At week 30, participants will stay in the clinic again and repeat the tests.

Participants will have a final visit 12 weeks after stopping treatment. This includes blood and urine tests.

...

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) and its progressive form, non-alcoholic steatohepatitis (NASH), are leading causes of liver injury and are tightly associated with obesity, diabetes and the metabolic syndrome. Despite recent advances, there is still a considerable knowledge gap regarding the fundamental pathogenic mechanisms, and especially regarding the transition from benign steatosis to steatohepatitis. Although NAFLD reflects disordered energy metabolism in the liver, little information exists on the response of the human liver to the acute caloric load of a meal. We hypothesize, based on preliminary non-invasive results, that in patients with NAFLD, an oral carbohydrate load results in preferential de novo lipogenesis (due to selective insulin resistance) and generation of fatty acids (FA). We further hypothesize a spillover effect, wherein NASH patients have an impairment of the hepatic ability to esterify the load of FA to triglycerides (TG) compared to patients with steatosis, resulting in accumulation of lipotoxic intermediary metabolites.

GLP-1 receptor agonists (GLP-1RA) have demonstrated significant benefit in the treatment of diabetes and obesity. Liraglutide was shown in a prospective trial to improve NASH histology and other GLP-1RA have shown benefit in secondary analyses, consistent with a class effect. However, response rates to GLP-1RA, as well as to other pharmacological interventions in NAFLD, have not exceeded 50%, and there are no adequate baseline predictors of response that could allow for selection of subjects for personalized treatment. Given that GLP-1RAs exert their main activity in the post-prandial state, it is plausible that post-prandial parameters may be more effective in predicting treatment response and can shed light on its mechanism.

Our aims in this study are (1) to assess the hepatic response to an acute oral carbohydrate load; (2) to identify which baseline parameters can predict the clinical response of NAFLD patients to a course of semaglutide, a novel GLP-1RA.

We propose a non-randomized, single-center, pilot exploratory study in which 32 subjects with steatosis (12-20) or NASH (12-20) will initially undergo two liver biopsies, one in the fasting state and one performed 2 hours after an oral 75g glucose load (OGTT biopsy). Tissue samples obtained will be subjected to a comparative, paired analysis of gene expression, protein phosphorylation in key signaling pathways, composition of tissue lipid species and oxidative stress. Subjects will be treated with semaglutide (escalated to 1 mg/week) for 30 weeks in all subjects, and their clinical response will be assessed by ALT and 1H-Magnetic resonance spectroscopy and a final (3rd) liver biopsy. Clinical responders will be compared to non-responders with regards to their baseline fasting and post-prandial parameters, to identify predictors of response.

The human hepatic response to a meal has never been studied at the tissue level and the findings of this study are likely to generate important data and clarify some of the fundamental questions regarding mechanisms of injury and insulin resistance. Furthermore, our study aims at identifying predictors of response to GLP-1RA and allow for appropriate selection of subjects for this class of medications, as well as to shed light on mechanism of response.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male or female Aged >= 18 years of age.
  2. Histological evidence of hepatic steatosis on a liver biopsy within 12 months OR evidence of fatty liver disease, as documented by imaging (ultrasound, CT, MRI, MRI-PDFF, MR spectroscopy, or Fibroscan CAP >= 285 db/M25) within 12 months.
  3. Estimated average alcohol consumption < 30 g/d for men or < 20 g/d for women in the 6 months prior to enrollment and no binge-drinking behavior.
  4. Ability of subject to understand and the willingness to sign a written informed consent document.

Additional Inclusion Criteria for Treatment Phase

1. Presence of NAFLD (steatosis grade greater than or equal to 1 on NASH-CRN scoring scale) on baseline admission liver biopsy.
2. Liver fat content greater than or equal to 10% by 1H-MRS on initial admission.

EXCLUSION CRITERIA:

1. Pregnant or breast-feeding
2. Chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV). Patients who were treated successfully for HCV and achieved sustained virological response can be eligible for enrollment > 18 months after treatment cessation. Patients receiving antiviral therapy are ineligible.
3. HIV infection.
4. Concomitant liver disease such as autoimmune hepatitis, primary biliary cholangitis, primary sclerosing cholangitis, Wilson s disease, alpha-1 antitrypsin deficiency, hereditary hemochromatosis.
5. Presence of definite or probable drug-induced liver injury. In the case of lipid-lowering, anti-hypertensive or anti-diabetic medications that are suspected to cause aminotransferase elevation, patients will be eligible if treatment is associated with stable enzyme levels for at least 6 months.
6. Decompensated advanced liver disease, defined as direct bilirubin > 0.5 g/dL, PT > 18 , albumin < 3 g/dL, MELD score > 12 (applicable only in patients without Gilbert s syndrome), or history of ascites, encephalopathy, variceal bleeding, spontaneous bacterial peritonitis or liver transplant
7. Treatment with medications known to cause fatty liver disease such as atypical neuroleptics, tetracycline, methotrexate or tamoxifen
8. Uncontrolled hypo- or hyperthyroidism.
9. Thyroid nodules with ultrasonographic features suggestive of an increased risk of thyroid cancer per radiologist reporting (hypoechoic, microcalcifications, twinkling on B flow imaging, central vascularity, irregular margins, incomplete halo, nodule taller than wide and documented enlargement of a nodule), or nodules associated with an abnormal TSH (0.4 to 5 mU/L).
10. Active coronary artery disease, defined as persistent angina pectoris, reversible ischemia on cardiac stress test or imaging, or the presence of significant coronary artery disease on imaging or catheterization. Patients with coronary artery disease that was treated by angioplasty or bypass surgery may be eligible if they have no evidence of active disease >= 1 year after intervention, can safely stop antiplatelet and anticoagulant medications before the performance of invasive procedures, and have adequate ventricular function as assessed by echocardiography or cardiology consultation. These patients will require cardiology consultation and clearance prior to enrollment.
11. Congestive heart failure.
12. Chronic kidney disease, with creatinine clearance < 60 ml/min or eGFR < 60/ml/min/m(2).
13. Uncontrolled diabetes mellitus with HbA1c > 9% will exclude subjects. Patients with diabetes may be enrolled only if they have HbA1c <=9%, have been on stable therapy with lifestyle and/or metformin for at least 3 months prior to enrollment, and are not foreseen to require change of antidiabetic medication or dose during the trial.
14. Use of insulin, sulfonylurea agents, thiazolidinediones, SGLT2 inhibitors, GLP-1 receptor agonists or DPP-4 inhibitors unless discontinued greater than or equal to 3 months before enrollment.
15. Contraindication or inability to perform a liver biopsy.

    1. Patients with coagulopathy (PT/PTT values that are prolonged greater than or equal to 3 seconds from the upper limit of the normal, including treatment with oral and parenteral anticoagulants), thrombocytopenia (< 70,000), abnormal bleeding time or platelet dysfunction. Antiplatelet agents taken for cardiovascular prevention will not exclude patients, unless they cannot be stopped safely for the performance of a liver biopsy.
    2. Hemoglobin level < 11 g/dL
16. Contraindications to MRI (heart pacemakers, unless MRI safe, insulin pumps, implanted hearing aids, neurostimulators, intracranial metal clips, metallic bodies in the eye, metal hip replacements, sutures, extreme anxiety or fear of small spaces.)
17. History of gastric bypass or other bariatric surgery, partial or complete gastrectomy and known maldigestion or malabsorption.
18. Treatment with orlistat.
19. Patients with uncontrolled eating disorders including anorexia and bulimia nervosa.
20. Patients with proliferative diabetic retinopathy.
21. Use of medications or supplements to treat NAFLD (approved or unapproved) unless withdrawn greater than or equal to 3 months prior to enrollment or taken at a stable dose for greater than or equal to 6 months.
22. Patients who had a liver biopsy performed less than or equal to 2 years before enrollment, unless they are willing to undergo all of the trial biopsies, knowing that these biopsies are purely for research and are not clinically indicated. This will be clearly documented in the patients charts prior to enrollment.
23. Inability or unwillingness to receive subcutaneous injections.
24. Known or suspected allergy to trial medication(s), excipients, or related products.
25. Alcohol or substance abuse within the past 12 months.
26. For women of childbearing potential, breast-feeding, pregnancy or inability or unwillingness to practice contraception for the duration of the study.
27. Personal or first-degree family member with history of medullary thyroid carcinoma or subjects with known multiple endocrine neoplasia syndrome type 2 (MEN-2).
28. Actively pursuing an intensive weight loss regiment, aimed at losing > 10% of current body weight, by following a different diet or exercise regimen over the study time period or recent (<3 months) significant weight loss (>10%).
29. The receipt of any investigational drug within 3 months prior to enrollment in this trial.
30. Assessment by the principal investigator that the subject will be unlikely to complete the study procedures, or that enrollment puts the subject at a significant risk unspecified by the criteria above.

INCLUSION CRITERIA for Healthy Volunteers (arm C)

1. Male or female Aged greater than or equal to 18 years of age.
2. No evidence of hepatic steatosis by imaging or histology.
3. No history of known liver disease.
4. Individuals on regular systemic medications may be considered eligible, and their eligibility will be determined by the principal investigator.
5. BMI less than or equal to 25 kg/m2
6. Non-diabetic.
7. Normal transaminases (ALT less than or equal to 31 U/L for men or less than or equal to 19 U/L for women, and AST less than or equal to 30 U/L).
8. Fasting glucose less than or equal to 95 mg/dL.
9. Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA for Healthy Volunteers (arm C)

1. Pregnant or breastfeeding
2. Excessive alcohol consumption, defined as an average alcohol consumption over > 1 drink per day over the past month
3. Assessment by the principal investigator that the subject is unsuitable for participation in the study or that enrollment puts the subject at significant risk.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-07-24 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Histological Improvement | 30 weeks
  >= point decrease in NAFLD activity score (range 0-8, high scores indicate more activity)
Clinical Improvement | 30 weeks
  Reduction of liver fat content (measure with 1H-magnetic resonance spectroscopy) by >= 25% and reduction of ALT by >=25% or normalization of ALT
Change in hepatic gene expression | 2 hours after an oral 75g glucose load
  Change in hepatic gene expression for biopsies performed at baseline and 2 hours after an oral 75g glucose load

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Rotman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
I will share human data generated in this research for future research as follows (check all that apply): @@@@@@@@@@@@_X_ De-identified data in an NIH-funded or approved public repository
Supporting Information: Study Protocol, ICF
Time Frame: IPD will shared at the time of publication or 6 months after publication.
Access Criteria: Data will be shared through: @@@@@@@@@@@@ An NIH-funded or approved public repository. Insert name or names: NIDDK repository or a similar database.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-DK-0072.html